CLINICAL TRIAL: NCT02979080
Title: The Evaluation of Iron Supplementation and Iron Requirements Using a Novel Isotope Dilution Method in Beninese Women
Brief Title: Iron Long-Term Labelling Study Benin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Michael B. Zimmermann (Other)
Responsible Party: Sponsor-Investigator, Prof. Michael B. Zimmermann, Professor, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Fe_LTL_Be
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Iron Absorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Iron Supplementation (Experimental): Eisensulfat LOMAPHARM 50 mg administration for 120 days
  Interventions: Other: Eisensulfat LOMAPHARM 50 mg

INTERVENTIONS:
Other: Eisensulfat LOMAPHARM 50 mg — Eisensulfat LOMAPHARM 50 mg administration for 120 days

SUMMARY:
Conventional indirect indicators of iron status, using serum and red blood cell biomarkers, are confounded by inflammation from common infections in sub-Saharan Africa, a region with a high prevalence of iron deficiency, making the assessment of iron balance and efficiency of iron intervention difficult. A potential reference method to quantify iron absorption and requirements using isotope dilution measurements in women living in areas with high burden of infection should be developed and validated within this project. The new method will allow accurate measurement of long term oral iron absorption and the estimation of iron requirements, potentially providing fundamental guidance for supplementation and fortification programs in sub-Saharan Africa. In a case series with four months' preventative iron supplementation intervention imbedded between a four months' control period prior intervention and a four months' control period after intervention, we will follow a group of 63 women. During the intervention period, the women will receive 50 mg Fe as ferrous sulfate tablets every day for 120 d. In total, the women will give 9 blood samples (day 1, 60 120, 150, 180, 210, 240, 300 and 360) for the de-termination of the isotopic composition and iron status biomarkers and 5 stool samples (day 1, 120, 180, 240 and 360) for the detection of soil transmitted helminths and gut inflammation. This design will allow the measurement of the isotopic iron dilution to assess the total oral iron absorption during the intervention period in comparison with the control periods without the administration of additional iron isotopes.

ELIGIBILITY:
Inclusion Criteria

* Have participated in one of the original absorption studies
* Signed written informed consent to participate in the study

Exclusion Criteria

* Long-term medication [except contraceptives]
* Any severe metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases according to the participants own statement or examination of study doctor
* Blood losses [surgery, accident], donations or transfusions during the past 4 months before study start.
* Residence too far away [1 hour or more by motorbike] from study locations; Natitingou or Cotonou

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
iron isotope composition in blood | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Benin (2):
  - Hôpital de zone de Natitingou, Natitingou, Atakora Department
  - Hôpital de zone d'Abomey-Calavi-Sô-Ava, Abomey-Calavi, Calavi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Speich C, Mitchikpe CES, Cercamondi CI, Zeder C, Brittenham GM, Moretti D, Zimmermann MB. Direct assessment of body iron balance in women with and without iron supplementation using a long-term isotope dilution method in Benin and Switzerland. Am J Clin Nutr. 2021 Jun 1;113(6):1657-1669. doi: 10.1093/ajcn/nqaa433. PMID 33693464